CLINICAL TRIAL: NCT06307340
Title: Adaption of the STAIR-NT Trauma Intervention for Polysubstance Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-01058
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Polysubstance Abuse; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Narrative Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analyst is blinded to participant arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted STAIR-NT Intervention (Experimental)
  Interventions: Behavioral: Skills Training in Affective and Interpersonal Regulation with Narrative Therapy (STAIR-NT)
- Treatment as Usual (TAU) (Active Comparator)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Skills Training in Affective and Interpersonal Regulation with Narrative Therapy (STAIR-NT) — Adapted version of evidence-based behavioral PTSD intervention.
  Arms: Adapted STAIR-NT Intervention
Behavioral: Treatment as Usual — Treatment as usual.
  Arms: Treatment as Usual (TAU)

SUMMARY:
During this 36-month R34 trial, eight study phases are proposed to adapt an evidence-based post traumatic stress disorder (PTSD) intervention (STAIR-NT) and layer it into a methadone maintenance treatment (MMT) program (START Treatment and Recovery centers) in New York City for use among individuals engaged in stimulant-opioid polysubstance use. The study aims to adapt STAIR-NT to a massed treatment schedule. Once an adapted protocol is complete, it will be tested for feasibility, acceptability, and short-term polysubstance and PTSD symptomology outcomes in a pilot randomized control trial (RCT) of 80 participants. Participants who screen eligible and consent will be randomized 1:1 to the adapted STAIR-NT intervention or treatment as usual (TAU) using randomization blocks of two and two and four via a computer-generated randomization sequence. Participants assigned to the intervention will receive the adapted massed delivery of STAIR-NT by trained counselors.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 years or older,
* be a patient at the START clinic receiving methadone for treatment of opioid use disorder,
* self-report 10+ days of co-use of cocaine and illicit opioids in the past 30-days,
* meet the criteria for stimulant use disorder (cocaine type; mild, moderate or severe) and a score of 3≥ on the PC-PTSD-5.

Exclusion Criteria:

* cognitive impairment that would interfere with their ability to understand study participation as assessed by the researcher,
* does not speak/understand English at a conversational level,
* plans to leave the START clinic in the next 60 days,
* patients who missed methadone doses (inactive) for 30 days or more, or
* having received clinical care from the interventionist(s) in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Eligible Participants | Baseline
  Proportion of persons eligible to enroll in the study of all possible MMT patients approached. Assessed using count data of individuals failing screen.
Proportion of Eligible Participants who Enroll | Baseline
  .Proportion of all eligible persons who enroll. Assessed using count data of individuals consented.
Number of Intervention Sessions Completed | Up to Month 3
Clinician-Rated Feasibility of Intervention Measure (FIM) Score | Month 3
  4-item, clinician-rated assessment of the feasibility of the intervention. Each item is rated on a scale from 1 (Completely disagree) to 5 (Completely agree); the total score is the sum of responses and ranges from 4-20. Higher scores indicate greater clinician-rated feasibility.
Clinician-Rated Feasibility of Acceptability of Intervention Measure (AIM) Score | Month 3
  4-item, clinician-rated assessment of the acceptability of the intervention. Each item is rated on a scale from 1 (Completely disagree) to 5 (Completely agree); the total score is the sum of responses and ranges from 4-20. Higher scores indicate greater clinician-rated acceptability.
Number of Days of Co-Use of Cocaine and Illicit Opioids | Month 3
  Measured using the Addiction Severity Index (ASI) questionnaire.
Number of Substances Used based on ASI Self-Report | Month 3
  Measured using the Addiction Severity Index (ASI) questionnaire, a self-report assessment to gauge the severity of a person's substance abuse.
Number of Substances Used based on Urine Drug Screen | Month 3
Number of Substances Used based on Chart Abstraction of Toxicology Results | Month 3
PTSD Checklist for DSM-5 (PCL-5) Score | Month 3
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Each item is rated on a scale from 0-4. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items; higher scores indicate greater severity of PTSD.
Negative Mood Regulation Scale Score | Month 3
  30-item assessment of individuals' beliefs and expectations regarding their ability to regulate their negative mood and emotions. Each item is rated on a 5-point Likert scale ranging from 1 (not at all effective) to 5 (extremely effective). The total score ranges from 30-150; higher scores indicate more effective negative mood regulation.
Inventory of Interpersonal Problems Score | Month 3
  A 127-item, self-report inventory that asks participants to rate a variety of interpersonal problems that may cause distress. The items are divided into two groups: (1) interpersonal inadequacies or inhibitions (78 items), (2) excesses or compulsions (49 items). Participants rate each item on a scale from 0 to 4 on how much difficulty/distress they feel regarding the item. The total score is calculated by adding the item responses; lower scores indicate less difficulty/distress.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Bunting, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Florida State University, Tallahassee, Florida
  - START Treatment and Recovery Centers, Brooklyn, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Deidentified quantitative assessment data will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research. Data will be stored in a data repository. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. The data will be stored in a data repository.

REFERENCES:
- [Derived] Renn T, Griffin B, Kumaravelu V, Ventuneac A, Santacatterina M, Bunting AM. Study protocol for a randomized controlled trial to adapt a posttraumatic stress disorder intervention of patients with opioid-stimulant polysubstance use receiving methadone maintenance treatment. BMC Psychiatry. 2024 Dec 4;24(1):879. doi: 10.1186/s12888-024-06348-0. PMID 39627789